CLINICAL TRIAL: NCT00658905
Title: A Prospective, Randomized, Double-blind Crossover Study Comparing 0.15 g/L rhBSSL Added to Infant Formula Versus Placebo During One Week of Treatment in Preterm Infants Born Before Week 32 of Gestational Age
Brief Title: Efficacy and Safety of Bile Salt Stimulated Lipase (BSSL) as Replacement Therapy in Infant Formula for Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BVT.BSSL-020
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Replacement Therapy in Preterm Infants
Keywords: Preterm infants; Replacement therapy; Infant formula; BSSL; BSSL is present in fresh mother's milk but not in infant formula.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBSSL (Active Comparator)
  Interventions: Drug: rhBSSL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhBSSL — 0.15 g/L rhBSSL added to infant formula; one week treatment
  Other Names: bucelipase alfa (INN)
  Arms: rhBSSL
Drug: Placebo — One week treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy in preterm infants following treatment with BSSL when administered in infant formula.

DETAILED DESCRIPTION:
In this double-blind crossover study, patients will be randomized to receive infant formula including BSSL or infant formula without BSSL for the first 7 days. After a wash-out period of 2 days the patients will "crossover" to the other treatment regimen and receive an additional 7 days treatment. The primary efficacy measurements will be made by collecting stool during the last three days of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants
* less than or equal to 32 weeks of gestational age
* appropriate for gestational age
* enterally fed with infant formula

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Coefficient of Fat Absorption in stool | Stool collected for a 72-hour period during the final 3 days of each treatment period

SECONDARY OUTCOMES:
Change in length and body weight between the start and end of each treatment period | Baseline and after one week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Timdahl, MD, Study Director — Biovitrum AB
Locations (6):
- Italy (6):
  - Presidio Ospedaliero di Alta Specializzazione G.Salesi Azienda Ospedaliero Universitaria Ospedali Riuniti "Umberto I-G.M.Lancisi -G.Salesi, Ancona
  - Azienda Ospedaliera "Ospedale Policlinico Consorziale",U.O Neonatologia e Terapia Intensiva Neonatale, Bari
  - 3) U.O. di Neonatologia e Terapia Intensiva Neonatale Università degli Studi di Milano, Ospedale Maggiore Policlinico,Mangiagalli e Regina Elena-Fondazione IRCCS, Milan
  - 4) Policlinico Universitario-Azienda Ospedaliera di Padova, Dipartimento di Pediatria, Padua
  - Clinical Pediatrica-Neonatologia, Policlinico Gemelli, Universita Cattolica, Rome
  - U.O. Neonatologia, Patologia Neonatale e Terapia Intensiva, Rome

REFERENCES:
- [Derived] Casper C, Carnielli VP, Hascoet JM, Lapillonne A, Maggio L, Timdahl K, Olsson B, Vagero M, Hernell O. rhBSSL improves growth and LCPUFA absorption in preterm infants fed formula or pasteurized breast milk. J Pediatr Gastroenterol Nutr. 2014 Jul;59(1):61-9. doi: 10.1097/MPG.0000000000000365. PMID 25222806